CLINICAL TRIAL: NCT04884295
Title: A 2-part Clinical Study Including a First in Human, Open Label, Single Ascending Dose Part (Phase 1) Followed by a Randomised, Double Blind, Placebo-controlled Part (Phase 2) to Evaluate the Efficacy and Safety of XVR011 in Patients Hospitalised for Mild to Moderate Coronavirus Disease 2019 (COVID-19)
Brief Title: Dose-Finding, Safety, and Efficacy Study of XVR011 Added to Standard of Care in Patients Hospitalised for COVID-19
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The sponsor does not intend to start Part 2 (Phase 2) due to change in company strategy for phase 2 design. This early end of trial is not due to reasons of safety or lack of efficacy. Part 1 (Phase 1) is completed as per protocol.
Sponsor: ExeVir Bio BV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EXEVIR0101; 2020-005299-36 (EudraCT Number)
Record Dates: First submitted 2021-05-06; First posted 2021-05-12 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — XVR011

STUDY DESIGN:
Intervention Model Description: Phase 1 is open-label, single ascending dose (completed per protocol); Phase 2 is double-blind, randomised, placebo-controlled (cancelled due to due to change in company strategy for phase II design)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- XVR011 (Experimental): Single Ascending Dose with 3 dose cohorts: low dose - medium dose - high dose (Phase 1)
  Interventions: Drug: XVR011

INTERVENTIONS:
Drug: XVR011 — Single dose of XVR011 via intravenous (IV) infusion

SUMMARY:
This is a 2 part study where the first part (Phase 1) evaluates the safety of XVR011 and aims to identify the recommended Phase 2 dose. The second part (Phase 2) follows after the part 1 and evaluates whether XVR011 added to standard of care in patients hospitalised for mild to moderate COVID-19 is a safe, well tolerated, and effective treatment.

Part 1 (Phase 1) is completed as per protocol. The sponsor does not intend to start Part 2 (Phase 2) due to change in company strategy for phase 2 design.

ELIGIBILITY:
Inclusion Criteria:

* Is ≥ 18 years of age.
* Tested positive for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) by RT-PCR and/or antigen test.
* Had an onset of COVID-19 symptom(s) within 8 days prior to screening; except for dyspnoea and/or tachypnoea for which an onset within 2 days prior to screening is applicable.
* Requires hospitalisation for medical care.
* Has oxygen saturation >= 91%.

Exclusion Criteria:

* Requires non-invasive or invasive mechanical ventilation and/or intensive care.
* Symptoms consistent with severe COVID-19.
* Has received a monoclonal antibody, plasma from a person who recovered from COVID-19 or any investigational treatment for COVID-19 within 30 days prior to study treatment.
* Has received an investigational or approved vaccination against SARS-CoV-2 within 14 days prior to study treatment.

NOTE: Other protocol defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2022-03-18 (Actual); Study Completion 2022-03-18 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with Adverse Events (all and serious) | Through Day 29
  Phase 1

SECONDARY OUTCOMES:
Total duration of oxygen supplementation | Through Day 29
  Phase 1
Proportion of subjects requiring mechanical ventilation and/or ICU transfer | Through Day 29
  Phase 1
Proportion of subjects with COVID-19 related symptoms | Through Day 29
  Phase 1
All-cause mortality rate | Through Day 29
  Phase 1
Change from baseline in the viral load (RT-qPCR) of nasopharyngeal samples | Up to Day 8/ Day of Discharge
  Phase 1
Time to recovery (i.e., clinical status reaching level 1 to 3 of the 8-point ordinal scale) | Through Day 29
  Phase 1
Time to hospital discharge | Through Day 29
  Phase 1

OTHER OUTCOMES:
Maximum serum concentration (Cmax) | Through Day 29
  Phase 1
Area under the serum concentration-time curve (AUC) | Through Day 29
  Phase 1
Serum terminal elimination half-life (t1/2) | Through Day 29
  Phase 1
Incidence of anti-drug antibody (ADA) to XVR011 | Through Day 29
  Phase 1

CONTACTS AND LOCATIONS:
Locations (6):
- Belgium (3):
  - Investigative Site, Ghent
  - Investigative Site, Liège
  - Investigative site, Mechelen
- Italy (2):
  - Investigative site, Milan
  - Investigative Site, Roma
- Investigative site, Chisinau, Moldova

IPD SHARING:
Plan to Share IPD: No